CLINICAL TRIAL: NCT00864877
Title: A Randomised, Prospective Clinical Investigation to Compare Post-Operative Fracture Healing and Complication Rate After the Fixation of Ankle Fractures Using the Inion OTPS FreedomPlate Biodegradable Fixation System Versus Conventional Metal Screws and Plates.
Brief Title: Comparison of Biodegradable & Metal Plates for Fixing Ankle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inion Oy (Industry)
Purpose: Treatment
Other Study IDs: D355 - 001
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Distal Fibular Fracture; Bimalleolar Fracture; Trimalleolar Fracture
Keywords: retrospective; comparison; biodegradable; implant; ankle fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: biodegradable fixation system (Inion OTPS FreedomPlateTM)
  Other Names: Inion OTPS(tm) FreedomPlate

SUMMARY:
A randomised, prospective clinical investigation to compare post-operative fracture healing and complication rate after the fixation of ankle fractures using the Inion OTPS FreedomPlateTM Biodegradable Fixation System versus conventional stainless steel metal screws and plates.

The objectives of the investigation are

* to compare post-operative fracture healing (union rates, time-to-union), and the complication rates (hardware failure, infection) between the two Plating Systems (biodegradable INION OTPS FreedomPlateTM vs. Stainless Steel 3.5 Reconstruction or DCP plate, or 1/3 Semitubular plates) at the clinical setting of Ankle fractures
* to study the safety of the clinical application of the biodegradable plating system of Inion OTPS FreedomPlateTM at the acute Ankle fracture setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to understand, sign and date the study-specific, Institutional Review Board/Ethics Committee approved patient informed consent and applicable privacy regulations.
2. Patient must require surgical treatment of a ankle fracture, with a distal fibular (i.e., lateral malleolus) fracture (isolated, closed, unilateral, non-comminuted) including either instable/dislocated Weber class B or any Weber class C fracture that cannot be anatomically reconstructed accurately without open procedure, or bimalleolar fracture with lateral malleolus fracture (as described above) and medial malleolus fracture (closed, unilateral, non-comminuted), or trimalleolar fracture with lateral and medial malleolus fractures as described above and posterior malleolus fracture with less than ¼ of the articular surface fractured
3. Fresh/acute fractures (seen within seventy-two hours of the injury)
4. Aged between 18 to 60 years
5. Skeletally mature
6. Willingness to accept randomisation either to the test or control group
7. Willingness and ability to comply with all investigation procedures pre- and post-operation.

Exclusion Criteria:

1. Contraindications of operative internal plate fixations
2. Contraindications for the Inion OTPS FreedomPlateTM Biodegradable Fixation System:

   * active or potential infection
   * patient's conditions, including limited blood supply, insufficient quantity or quality of bone, and where patient cooperation cannot be guaranteed (e.g., alcoholism, drug abuse)
   * high-load bearing applications
3. Multiple trauma, head injury, bilateral lower extremity fractures, upper extremity fractures
4. Any concomitant painful or disabling disease of the lower limb that would interfere with evaluation of the affected ankle
5. Previous ankle fracture
6. Patients who most likely will not learn to walk with crutches (e.g., due to being severely overweight)
7. Bone malignancy
8. Osteomyelitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2009-05; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The functional performance will be primarily determined by the Olerud and Molander Ankle Score | at 2, 6 and 12 weeks, and 12 and 24 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, Professor, Principal Investigator — Leeds General Infirmary
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom